CLINICAL TRIAL: NCT00135837
Title: An Open-Label, Multicenter, Phase 4 Study of the Effect of Verteporfin for Injection Therapy in Subjects With Occult With No Classic Choroidal NeoVascularization Secondary to Age-Related Macular Degeneration
Brief Title: Photodynamic Therapy in Occult-Only Lesions (POOL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: QLT Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBPD952B2401
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2006-06-21 (Estimated); Status verified 2006-06

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age related Macula Degeneration,; AMD,; choroidal neovascularisation (CNV),; occult CNV lesion,; verteporfin for injection,; photodynamic therapy (PDT)
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Verteporfin; Injections

INTERVENTIONS:
Drug: Verteporfin for injection

SUMMARY:
Age related macular degeneration is the leading cause of blindness for people over 50 in the western world. Blood vessels which start to grow form a lesion in the back of the eye. Verteporfin may stabilize the disease, by closing the blood vessels. This study will assess the efficacy and safety of verteporfin in patients with occult only lesions.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older
* Must see better or equal to 34 letters (visual acuity)
* Choroidal neovascularization (CNV) lesion must be occult only

Exclusion Criteria:

* Evidence of classic CNV in the lesion
* Prior treatment of disease in study eye
* Have a history of moderate to severe hepatic impairment

Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202
Dates: Start 2003-06

PRIMARY OUTCOMES:
visual acuity measurements, baseline, 12 months

SECONDARY OUTCOMES:
visual acuity measurements, fundus photographs and fluorescein angiography at baseline, 12 months; ophthalmic examinations, adverse events, vital signs, concomitant medications, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Customer Information, Study Chair — Novartis
Locations (1):
- Novartis, Basel, Switzerland